CLINICAL TRIAL: NCT02155985
Title: Modulation of Immune Activation by Aspirin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5331; UM1AI068636 (NIH)
Record Dates: First submitted 2014-06-03; First posted 2014-06-04 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aspirin 300 mg + aspirin 100 mg placebo (Active Comparator): At week 0, participants were prescribed aspirin 300 mg (one tablet) and placebo for aspirin 100 mg (one tablet) once daily. At week 12, participants were to stop both study product tablets to allow for a 4-week washout period.
  Interventions: Drug: Aspirin; Drug: Placebo
- Aspirin 100 mg + aspirin 300 mg placebo (Active Comparator): At week 0, participants were prescribed a placebo for aspirin 300 mg (one tablet) and aspirin 100 mg (one tablet) once daily. At week 12, participants were to stop both study product tablets to allow for a 4-week washout period.
  Interventions: Drug: Aspirin; Drug: Placebo
- Aspirin 300 mg + aspirin 100 mg placebos (Placebo Comparator): At week 0, participants were prescribed a placebo for aspirin 300 mg (one tablet) and placebo for aspirin 100 mg (one tablet) once daily. At week 12, participants were to stop both study products tablets to allow for a 4-week washout period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Aspirin is a nonsteroidal antiinflammatory drug (NSAID) effective in treating fever, pain, and inflammation in the body.
  Arms: Aspirin 100 mg + aspirin 300 mg placebo; Aspirin 300 mg + aspirin 100 mg placebo
Drug: Placebo — Placebo for aspirin

SUMMARY:
Since people started taking HIV medications, illness from AIDS has decreased, but other serious diseases like heart disease, cancer, and kidney, and liver disease have increased. HIV causes inflammation (irritation) inside the body that cannot be felt but can be measured by blood. Inflammation can lead to diseases that have become some of the leading causes of death in people with HIV. HIV therapy can partially lower levels of inflammation measured in blood, however, levels of inflammation in people who have HIV may remain high compared with people not infected with HIV.

Aspirin is a drug that is commonly used for pain relief but is also approved by the Food and Drug Administration (FDA) for preventing heart attacks and stroke in those who are at increased risk for heart attack and stroke. Aspirin also is used (but is not approved by the FDA) to decrease the risk of some cancers in people who are at increased risk. Aspirin is thought to decrease risk of heart attack and stroke because it blocks the activation of platelets and prevents blood clots from clogging narrowed blood vessels, a disease called atherosclerosis. It is unknown how aspirin might decrease the chance of developing cancer in some people at higher risk, but aspirin has been shown to modulate (or change) the immune system. In HIV-infected people who have been taking antiretroviral therapy and have an undetectable HIV viral load it was recently shown that low-dose aspirin 81 mg (baby aspirin), given for one week, lowers platelet activation and reduces blood markers of inflammation which may improve the function of the immune system.

The purpose of this study was to evaluate whether aspirin improves inflammation and immune activation when compared to a placebo (inactive medication like a dummy pill) and to determine if 12 weeks of aspirin 300 mg and aspirin 100 mg is safe for HIV-infected persons on antiretroviral therapy. Additionally, it studied whether a higher dose and longer duration of aspirin provides further anti-inflammatory and immune-modulating benefit. This was done using blood and urine tests that measure inflammation and also with a test that uses ultrasound to measure the flow of blood in your arm, called flow-mediated vasodilation (FMD) of the brachial artery (BART). This is a painless test that bounces sound waves off of a blood vessel in your arm.

DETAILED DESCRIPTION:
This was a phase II prospective, double-blind, randomized, placebo-controlled 3-arm clinical trial to study whether aspirin improves inflammation and immune activation. At study entry, participants were randomized between the three study arms: aspirin 300 mg, aspirin 100 mg and placebo. The study treatment duration was 12 weeks, followed by a 4 week washout period. The study duration was 16 weeks.

The study clinic visits included pre-entry (within 7 days prior to entry), entry, on treatment visits at weeks 2, 11 and 12, and final study visit at the end of the wash-out period at week 16. The samples for the primary and secondary outcomes were collected at pre-entry, entry, and weeks 2, 11 and 12. The evaluations of safety (clinical assessment for signs and symptoms, diagnoses, laboratory tests) were done at entry and weeks 2, 11, 12 and 16.

The co-primary objectives used pair-wise comparisons to assess the effects of 300 mg and 100 mg of daily aspirin for 12 weeks on plasma sCD14 levels.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection.
* Currently on continuous ART for ≥48 weeks prior to study entry. NOTE: This is defined as continuous active therapy with no treatment interruption longer than 7 consecutive days and a total duration off-treatment of no more than 14 days during the 48 weeks prior to entry.
* No change in ART regimen within the 12 weeks prior to study entry (except as noted below).

NOTE: Modifications of ART dosing during within the 12 weeks prior to entry are permitted. In addition, the change in formulation (eg, from standard formulation to fixed dose combination or single tablet regimen) or dosing (eg, from once a day to twice a day) is allowed within 12 weeks prior to entry. Within-class single drug substitution (eg, switch from nevirapine to efavirenz or from atazanavir to darunavir), are not allowed within 12 weeks prior to entry. No other changes in ART in the 12 weeks prior to entry are permitted.

* Screening HIV-1 RNA must be <50 copies/mL and performed by any FDA-approved assay at any US laboratory that has a CLIA certification or its equivalent within 45 days prior to study entry.
* Maintain ART-mediated viral suppression for at least 48 weeks prior to study entry defined as:

A. At least one HIV-1 RNA test result obtained at any time point greater than 48 weeks prior to study entry must be BLQ and must be performed by any FDA-approved assay at a CLIA-certified laboratory or its equivalent.

AND

B. All HIV-1 RNA tests reported during the 48 weeks prior to study entry must be BLQ and must be performed by any FDA-approved assay at a CLIA-certified laboratory or its equivalent.

NOTE: A single RNA "blip" of ≤500 copies/mL is permissible if RNA levels most recent before and after (may include the screening HIV-1 RNA test) are below the level of quantification (BLQ) for the assay. If the RNA level after the blip is the screening HIV-1 RNA test, the result must be <50 copies/mL.

* The following laboratory values obtained within 45 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent.

  * Absolute neutrophil count (ANC) ≥750/mm^3
  * Hemoglobin ≥9.0 g/dL for female subjects and ≥10.0 g/dL for male subjects
  * Platelet count >100,000/mm^3
  * Prothrombin time (PT) <1.2 x upper limit normal (ULN)
  * Partial thromboplastin time (PTT) <1.5 x ULN
  * Calculated creatinine clearance (CrCl) ≥30 mL/min, as estimated by the Cockroft-Gault formula NOTE: Calculation for the Cockcroft-Gault equation is available at https://www.fstrf.org/apps/cfmx/apps/common/Portal/index.cfm
  * Aspartate aminotransferase (AST) (SGOT) ≤2 x ULN.
  * Alanine aminotransferase (ALT) (SGPT) ≤2 x ULN.
  * Alkaline phosphatase ≤2 x ULN.
  * Total bilirubin ≤2.5 x ULN. If the subject if taking an indinavir- or atazanavir-containing regimen at the time of screening, a total bilirubin of ≤5 x ULN is acceptable.
* Female study volunteers of reproductive potential (pre-menopausal women who have not had a sterilization procedure (eg, hysterectomy, bilateral oophorectomy, tubal ligation, or salpingectomy) must have a negative serum or urine pregnancy test performed within 24 hours prior to study entry. Women are considered menopausal if they have not had a menses for at least 12 months and have a FSH (follicle stimulating hormone) of greater than 40 IU/L or, if FSH testing is not available, they have had amenorrhea for 24 consecutive months.

If the female volunteer is not of reproductive potential (women who are menopausal, defined as not having had a menses for at least 12 months with an FSH of greater than 40 IU/L, or if FSH testing is not available, have had amenorrhea for 24 consecutive months, or women who have undergone surgical sterilization, (eg, hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy)), she is eligible without requiring the use of a contraceptive method. Acceptable documentation of sterilization is subject reported history of hysterectomy, bilateral oophorectomy, tubal ligation, tubal micro-insert, menopause, or the partner with vasectomy/azoospermia.

- If participating in sexual activity that could lead to pregnancy, the female study volunteer must be willing to use contraception while receiving protocol-specified medication(s) and for the washout period of 4 weeks. At least one of the following methods MUST be used:

* Condoms (male or female), with or without a spermicidal agent
* Diaphragm or cervical cap with spermicide
* Intrauterine device (IUD)
* Hormone-based contraceptive

As hormone-based contraceptives (oral, transdermal, or subdermal) can affect coagulopathy biomarkers, subjects who plan on using such a contraceptive during the study must be taking the same product for ≥4 weeks prior to screening and be encouraged to continue throughout the duration of the study, if medically feasible.

* No documented opportunistic infections within 24 weeks prior to study entry
* Karnofsky performance score >/= 70 within 45 days prior to study entry
* Ability and willingness of subject or legal guardian/representative to provide written informed consent.
* Willingness to refrain from the use of aspirin or any aspirin-related product (other than the study drug), including NSAIDs, from time of screening visit through the end of the 16 week trial.

NOTE: Acetaminophen-based products may be used before and during the trial when analgesics are required.

* Completion of the pre-entry FMD assessment NOTE: The FMD must be performed at the site and confirmed as acceptable by the University of Wisconsin Atherosclerosis Imaging Research Program (UW AIRP) core lab prior to study entry.
* Confirmation of the availability of the stored pre-entry fasting specimens (plasma and serum); the site must confirm that these specimens have been entered into the Laboratory Data Management System (LDMS).

Exclusion Criteria:

- Current malignancy (except non-melanoma cancer of the skin not requiring systemic chemotherapy or radiation therapy).

NOTE: Carcinoma in situ of the cervix or anus is not considered exclusionary.

* Prior history of malignancy if the subject is not disease free for 24 or more weeks prior to study entry.
* Current use or indication for use of non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin that cannot be interrupted for clinical reasons. Examples of clinical reasons include, but are not limited to, known and documented cardiovascular disease (history of MI, coronary artery bypass graft surgery, percutaneous coronary intervention, stroke, transient ischemic attack, peripheral arterial disease with ABI <0.9 or claudication).
* Current diagnosis of diabetes with HbA1c ≥8% within 24 weeks prior to screening.
* Changes in lipid-lowering or antihypertensive medication within 90 days prior to study entry or expected need to modify these medications during the study.

NOTE: Lipid-lowering medication includes: statins, fibrates, niacin (dose ≥250 mg daily), and fish-oil/omega 3 fatty acids (dose >1000 mg of marine oils daily).

* Known cirrhosis
* Known chronic active hepatitis B NOTE: Active hepatitis B is defined as hepatitis B surface antigen positive and hepatitis B DNA positive within 24 weeks prior to study entry; subjects with hepatitis B virus (HBV) DNA BLQ for greater than 24 weeks prior to study entry are eligible.
* Known chronic active hepatitis C NOTE: Active hepatitis C is defined as a detectable plasma HCV RNA level within 24 weeks prior to study entry; subjects with HCV RNA BLQ for greater than 24 weeks prior to study entry are eligible.
* Known inflammatory conditions, such as, but not limited to, rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), sarcoidosis, inflammatory bowel disease (IBD), chronic pancreatitis, autoimmune hepatitis, Adult Stills disease, Rheumatic heart disease, bursitis.
* Breastfeeding or pregnant
* Previous intolerance or allergy to aspirin or any aspirin products.
* Frequent use of aspirin or aspirin products (NSAIDs), defined as an average of 2 or more times per week in the last 12 weeks prior to study entry.
* Immunosuppressant use, such as, but not limited to, systemic or potentially systemic glucocorticoids (including injected, ie, intra-articular, nasal or inhaled steroids), azathioprine, tacrolimus, mycophenolate, sirolimus, rapamycin, methotrexate, or cyclosporine within 45 days prior to study entry.
* Use of any systemic antineoplastic or immunomodulatory treatment, investigational vaccines, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 45 days prior to study entry.

NOTE: Routine standard of care, including hepatitis A and/or B, human papilloma virus, influenza, pneumococcal, and tetanus vaccines are permitted if administered at least 7 days before study entry and before biomarker/peripheral blood mononuclear cell (PBMC) blood collections.

* Concurrent use of prohibited medications as per section 5.4
* Heavy alcohol use as defined by the National Institute on Alcohol Abuse and Alcoholism (NIAAA) http://www.niaaa.nih.gov/alcohol-health/overview-alcohol-consumption/moderate-binge-drinking
* Alcohol or drug use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Current use of anticoagulation therapy or conditions requiring use of anticoagulants, use such as, but not limited to warfarin (Coumadin), rivaroxaban (Xarelto), clopidogrel (Plavix), dabigatran (Pradaxa), apixaban (Eliquis), heparin, ticlopidine (Ticlid), Presugrel (Effient).
* History of coagulopathy, deep venous thrombosis, pulmonary embolism.
* Known active or recent (not fully resolved within 4 weeks prior to study entry) invasive bacterial, fungal, parasitic, or viral infections.

NOTE: Recurrent herpes simplex virus (HSV) is not exclusionary. Subjects on antiviral prophylaxis for HSV or VZV are encouraged to remain on treatment for the duration of the study if medically feasible.

* Serious illness or trauma requiring systemic treatment and/or hospitalization within 4 weeks prior to study entry.
* History of bleeding conditions such as peptic ulcer disease, hemophilia, von Willebrand disease, idiopathic thrombocytopenic purpura.
* History of thrombotic disorders such as protein C or S deficiency.
* History of gastrointestinal (GI) bleeding within the past 6 months prior to study entry.
* History of intracranial hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Aberg, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Meagan O'Brien, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (15):
- United States (15):
  - 601 University of California, Los Angeles CARE Center CRS, Los Angeles, California
  - 701 University of California, San Diego AntiViral Research Center CRS, San Diego, California
  - Ucsf Aids Crs (801), San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - 2701 Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - 3201 Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - 3652 Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Houston AIDS Research Team CRS (31473), Houston, Texas

REFERENCES:
- See also: Version 2.0 of the DAIDS EAE Manual — http://rsc.tech-res.com/clinical-research-sites/safety-reporting/manual
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009), — http://rsc.tech-res.com/clinical-research-sites/safety-reporting/daids-grading-tables

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant enrolled on August 18, 2014. The last participant enrolled on March 6, 2015.
Pre-assignment Details: Participants were randomized to the three study arms using a 1:1:1 allocation ratio with permuted blocks of size 6 and without institutional balancing. There was no stratification.
Groups:
- Aspirin 300 mg + Aspirin 100 mg Placebo: At week 0, participants were prescribed aspirin 300 mg (one tablet) and placebo for aspirin 100 mg (one tablet) once daily. At week 12, participants were to stop both study product tablets to allow for a 4-week washout period.
  Aspirin
  Placebo for aspirin
- Aspirin 100 mg + Aspirin 300 mg Placebo: At week 0, participants were prescribed a placebo for aspirin 300 mg (one tablet) and aspirin 100 mg (one tablet) once daily. At week 12, participants were to stop both study product tablets to allow for a 4-week washout period.
  Aspirin
  Placebo for aspirin
- Aspirin 300 mg + Aspirin 100 mg Placebos: At week 0, participants were prescribed a placebo for aspirin 300 mg (one tablet) and placebo for aspirin 100 mg (one tablet) once daily. At week 12, participants were to stop both study products tablets to allow for a 4-week washout period.
  Placebo for aspirin
Period: Overall Study
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Started | 40 | 41 | 40
Completed | 39 | 41 | 39
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 121 randomized participants, all of which did initiate study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos | Total
Number analyzed (Participants) | 40 | 41 | 40 | 121
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [38 to 54] | 50 [46 to 56] | 49 [42 to 57] | 49 [42 to 55]
Age, Customized [Number; unit: participants]
  20 - 29 years | 5 | 1 | 1 | 7
  30 - 39 years | 7 | 5 | 7 | 19
  40 - 49 years | 10 | 12 | 13 | 35
  50 - 59 years | 15 | 18 | 13 | 46
  60 - 69 years | 3 | 4 | 5 | 12
  70 - 79 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 5 | 23
  Male | 32 | 31 | 35 | 98
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 21 | 18 | 21 | 60
  Black Non-Hispanic | 11 | 19 | 11 | 41
  Hispanic (Regardless of Race) | 7 | 4 | 8 | 19
  Asian, Pacific Islander | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 40 | 121
Smoking Status [Number; unit: participants]
  Never | 19 | 25 | 26 | 70
  Previously | 11 | 7 | 6 | 24
  Currently | 10 | 9 | 8 | 27
Statin Use [Number; unit: participants]
  Off Statins | 33 | 35 | 34 | 102
  Pravastatin | 3 | 0 | 3 | 6
  Atorvastatin | 3 | 5 | 3 | 11
  Rosuvastatin | 1 | 1 | 0 | 2
BMI, Continuous [Median (Inter-Quartile Range); unit: kg/m^2] | 25.9 [23.5 to 28.1] | 25.8 [22.8 to 30.2] | 27.3 [23.7 to 30.1] | 26.0 [23.4 to 29.2]
CD4 Count, Continuous [Median (Inter-Quartile Range); unit: cells/mm^3] | 573 [436 to 684] | 629 [481 to 856] | 642 [436 to 747] | 599 [456 to 777]
HIV-1 RNA, Categorical [Number; unit: participants]
  <40 copies/mL | 40 | 38 | 40 | 118
  41 copies/mL | 0 | 1 | 0 | 1
  45 copies/mL | 0 | 1 | 0 | 1
  162 copies/mL | 0 | 1 | 0 | 1
Platelets, Continuous [Median (Inter-Quartile Range); unit: 10^9/L] | 222.5 [192 to 251] | 229 [200 to 271] | 224.5 [184 to 258.5] | 226 [192 to 261]
Hemoglobin, Continuous [Median (Inter-Quartile Range); unit: g/dL] | 14.2 [13.4 to 15.0] | 14.1 [13.6 to 15.0] | 14.2 [13.4 to 15.4] | 14.2 [13.4 to 15.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in sCD14 From Baseline to Week 11/12
Description: Baseline is defined as the average of the Pre-Entry and Entry values. Week 11/12 is defined as the average of the Week 11 and Week 12 values. All values were log10 transformed prior to calculating change and conducting analyses. Values obtained within 6 days after the influenza vaccination were excluded.
  Absolute change was calculated as the value at week 11/12 minus the value at baseline. Mean changes were exponentiated to be back on the untransformed scale and corresponds to a mean fold change. Differences between arms are expressed as the percent difference between mean fold changes.
Time Frame: Pre-entry and entry to weeks 11 and 12
Population: Analysis used the per-protocol population. Participants 1) without baseline AND week 11/12 sCD14 values, or 2) with premature discontinuation of study treatment, or 3) with a serious bacterial infection while on treatment, or 4) with <70% self-reported adherence (based on all available days of recall) to study treatment were excluded.
Measure: Mean (95% Confidence Interval); unit: fold change
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 38 | 38 | 36
fold change | 0.99 [0.94 to 1.04] | 1.03 [0.98 to 1.08] | 0.97 [0.93 to 1.02]
Statistical Analysis 1: Comparison: Aspirin 300 mg + Aspirin 100 mg Placebo vs Aspirin 300 mg + Aspirin 100 mg Placebos; Paired differences between the two aspirin arms and placebo were estimated in a single linear regression model using linear combinations of the estimated means; Test type: Superiority or Other; p = 0.70, t-test, 2 sided — While there are co-primary comparisons, due to the pilot nature of the study, no adjustment to the 0.05 type I error was made; Mean Difference (Net) = 1.4, 95% CI 2-sided [-5.5 to 8.8] — Mean difference is the percent difference in mean fold changes = ((300 mg mean fold change / placebo mean fold change) - 1) * 100
Statistical Analysis 2: Comparison: Aspirin 100 mg + Aspirin 300 mg Placebo vs Aspirin 300 mg + Aspirin 100 mg Placebos; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.14, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 5.5, 95% CI 2-sided [-1.7 to 13.3] — Mean difference is the percent difference in mean fold changes = ((100 mg mean fold change / placebo mean fold change) - 1) * 100

2. Secondary Outcome: Safety
Description: Safety was summarized as the highest grade sign/symptom, laboratory event, or diagnosis per participant.
  Grading (Grade 0: normal, Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening) was done by site clinicians using DAIDS AE Grading table.
Time Frame: After study entry to Week 16
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 40 | 41 | 40
Participants
  Grade 0 | 37 | 37 | 33
  Grade 1 | 1 | 1 | 1
  Grade 2 | 2 | 2 | 4
  Grade 3 | 0 | 1 | 2

3. Secondary Outcome: Tolerability
Description: Tolerability was summarized as the number of participants successfully completing the protocol-defined treatment period.
Time Frame: Treatment dispensation to Week 12
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 40 | 41 | 40
Participants | 38 | 40 | 38

4. Secondary Outcome: Change in sCD163 From Baseline to Week 11/12
Description: Baseline is defined as the average of the Pre-Entry and Entry values. Week 11/12 is defined as the average of the Week 11 and Week 12 values. All values were log10 transformed prior to calculating change and conducting analyses. Values obtained within 6 days after the influenza vaccination were excluded.
  Absolute change was calculated as the value at week 11/12 minus the value at baseline. Mean changes were exponentiated to be back on the untransformed scale and corresponds to a mean fold change.
Time Frame: Pre-entry and entry to weeks 11 and 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: fold change
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 38 | 38 | 36
fold change | 1.12 [1.03 to 1.23] | 1.03 [0.94 to 1.13] | 0.98 [0.89 to 1.07]

5. Secondary Outcome: Change in Expression of CD14dimCD16+ From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percentage of CD14dimCD16+
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percentage of CD14dimCD16+ | 0.13 [-0.88 to 1.14] | 0.27 [-0.74 to 1.28] | 0.15 [-0.86 to 1.16]

6. Secondary Outcome: Change in Expression of CD69+ on CD14dimCD16+ From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percent of CD14dimCD16+ expressing CD69+
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percent of CD14dimCD16+ expressing CD69+ | -0.12 [-4.52 to 4.29] | -2.22 [-6.62 to 2.19] | 1.82 [-2.58 to 6.23]

7. Secondary Outcome: Change in Expression of CD14+CD16- From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percentage of CD14+CD16-
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percentage of CD14+CD16- | 7.71 [1.52 to 13.89] | -0.48 [-6.66 to 5.71] | 2.62 [-3.56 to 8.81]

8. Secondary Outcome: Change in Expression of CD69+ on CD14+CD16- From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percent of CD14+CD16- expressing CD69+
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percent of CD14+CD16- expressing CD69+ | 4.16 [-2.18 to 10.49] | -0.27 [-6.60 to 6.07] | 3.33 [-3.01 to 9.66]

9. Secondary Outcome: Change in Expression of CD14+CD16+ From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percentage of CD14+CD16+
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percentage of CD14+CD16+ | -7.86 [-14.24 to -1.47] | 0.19 [-6.19 to 6.58] | -2.88 [-9.26 to 3.51]

10. Secondary Outcome: Change in Expression of CD69+ on CD14+CD16+ From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percent of CD14+CD16+ expressing CD69+
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percent of CD14+CD16+ expressing CD69+ | 1.07 [-5.29 to 7.43] | -3.48 [-9.83 to 2.88] | 2.12 [-4.24 to 8.48]

11. Secondary Outcome: Change in Expression of CD38+HLA-DR+ on CD4+ From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percent of CD4+ expressing CD38+HLA-DR+
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percent of CD4+ expressing CD38+HLA-DR+ | -1.46 [-2.98 to 0.05] | -0.94 [-2.45 to 0.58] | -0.03 [-1.56 to 1.51]

12. Secondary Outcome: Change in Expression of CD38+HLA-DR+ on CD8+ From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percent of CD8+ expressing CD38+HLA-DR+
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percent of CD8+ expressing CD38+HLA-DR+ | -1.16 [-2.85 to 0.54] | -1.47 [-3.17 to 0.23] | -0.48 [-2.21 to 1.24]

13. Secondary Outcome: Change in Expression of PD-1+ on CD4+ From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ expressing PD-1+
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percentage of CD4+ expressing PD-1+ | -0.46 [-1.81 to 0.88] | -0.19 [-1.53 to 1.16] | -0.75 [-2.11 to 0.62]

14. Secondary Outcome: Change in Expression of PD-1+ on CD8+ From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percentage of CD8+ expressing PD-1+
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 35 | 35 | 33
percentage of CD8+ expressing PD-1+ | -0.18 [-1.54 to 1.18] | -0.07 [-1.44 to 1.29] | -0.74 [-2.13 to 0.64]

15. Secondary Outcome: Change in IL-6 From Baseline to Week 11/12
Description: as for outcome 4
Time Frame: Pre-entry and entry to weeks 11 and 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: fold change
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 38 | 38 | 36
fold change | 1.03 [0.87 to 1.21] | 1.13 [0.96 to 1.33] | 0.92 [0.78 to 1.09]

16. Secondary Outcome: Change in D-dimer From Baseline to Week 11/12
Description: as for outcome 4
Time Frame: Pre-entry and entry to weeks 11 and 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: fold change
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 38 | 38 | 35
fold change | 1.08 [0.97 to 1.19] | 0.99 [0.89 to 1.10] | 1.02 [0.91 to 1.13]

17. Secondary Outcome: Change in Kynurenine to Tryptophan Ratio From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: 1000 ng/ml kynurenine : ng/ml tryptophan
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 38 | 37 | 35
1000 ng/ml kynurenine : ng/ml tryptophan | 0.45 [-1.78 to 2.69] | -2.60 [-4.90 to -0.30] | -1.26 [-3.59 to 1.07]

18. Secondary Outcome: Change in Serum Thromboxane B2 From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: fold change
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 38 | 36 | 33
fold change | 0.28 [0.20 to 0.38] | 0.20 [0.15 to 0.28] | 1.21 [0.86 to 1.69]

19. Secondary Outcome: Change in Urine Thromboxane Per Creatinine From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: fold change
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 38 | 37 | 33
fold change | 0.25 [0.19 to 0.32] | 0.23 [0.18 to 0.30] | 0.96 [0.71 to 1.30]

20. Secondary Outcome: Change in Brachial Artery Flow-mediated Dilation (FMD) From Entry to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at entry.
Time Frame: Entry to Week 12
Population: Analysis used the per-protocol population as in the primary analyses.
Measure: Mean (95% Confidence Interval); unit: percentage of brachial artery diameter
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
Number analyzed (Participants) | 34 | 33 | 32
percentage of brachial artery diameter | -0.32 [-1.17 to 0.54] | -0.98 [-1.85 to -0.11] | -0.20 [-1.08 to 0.69]

ADVERSE EVENTS:
Time Frame: From baseline to Week 16.
Description: Protocol required reporting: post-entry signs/symptoms >=Grade 3, laboratory results >=Grade 2, new diagnoses and events that led to a change in treatment, regardless of grade. The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (V1.0, December 2004 (Clarification, August, 2009)) and Expedited AE Manual (V2.0) were used.
Arm/Group | Aspirin 300 mg + Aspirin 100 mg Placebo | Aspirin 100 mg + Aspirin 300 mg Placebo | Aspirin 300 mg + Aspirin 100 mg Placebos
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 1/41 | 6/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin 300 mg + Aspirin 100 mg Placebo (N=40) | Aspirin 100 mg + Aspirin 300 mg Placebo (N=41) | Aspirin 300 mg + Aspirin 100 mg Placebos (N=40)
Acute sinusitis (Infections and infestations) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less